CLINICAL TRIAL: NCT03976050
Title: A Phase I, Single Arm, Dose Escalation Study to Evaluate Safety, Pharmacokinetics and Preliminary Efficacy of HL-085 in Subjects With Advanced Solid Tumors
Brief Title: Phase I Study of HL-085 in Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study objective and design change
Sponsor: Shanghai Kechow Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HL-085-US-101
Record Dates: First submitted 2019-06-02; First posted 2019-06-05 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Solid Tumor, Adult

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose escalation (Experimental): Subjects in the dose escalation cohorts will receive ascending doses of HL-085 until the MTD is determined. The first three subjects will receive twice-daily doses (BID) of HL-085 6 mg. Additional cohorts may receive doses of HL-085 9, 12 or 18 mg BID respectively and sequentially. If DLTs are observed in <33.3% of subjects at the 18 mg dose.
  Interventions: Drug: HL-085

INTERVENTIONS:
Drug: HL-085 — HL-085 is a MEK inhibitor with potential indication for cancers. it will be given twice daily continuously in the study until disease progression; or the risks outweigh the benefits, if the subject continues study treatment; or subjects with poor compliance; or subjects need to receive or have already started alternative anti-tumor drugs; or Subjects who need to receive or have already started alternative any other concomitant medication and/or treatment, which would significantly impact their safety; or interruption of IP administration for more than 14 days due to IP-related AEs.
  Other Names: No other interventions

SUMMARY:
The study drug, HL-085 is a MEK inhibitor with the potential indication for cancers. It is an oral medication to be given daily.

The purposes of this study is to find answers to the following research questions:

1. What is the highest tolerable dose of HL-085 that can be given to subjects when given orally (by mouth) on a twice daily basis?
2. What are the side effects of HL-085?
3. How much HL-085 is in the blood at specific times after dosing and how does the body get rid of the HL-085?

ELIGIBILITY:
Inclusion Criteria:

1. Must have a pathologically documented solid tumor(s) that has relapsed from, or is refractory to standard treatment, or for which no standard treatment is available.
2. Must have at least one measurable lesion as defined by RECISTv1.1 criteria for solid tumors.
3. Must have received biological chemotherapy, immunotherapy or radiotherapy ≥4 weeks prior to starting the study treatment. Must have received small molecule chemotherapy ≥2 weeks or five half-lives (whichever is longer) prior to starting the study treatment.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
5. Life expectancy ≥3 months (as judged by the Investigator).
6. Must have adequate hematologic, hepatic and renal function.

Exclusion Criteria:

1. Have undergone or plan to have major surgery or experienced severe trauma ≤28 days prior to starting the study treatment.
2. Known hypersensitivity to IP ingredients or their analogues.
3. Prior therapy with a MEK-inhibitor
4. Receipt of any other investigational agent therapy within 4 weeks prior to starting study treatment.
5. Any concurrent therapy for cancer treatment.
6. Have active central nervous system lesion.
7. Receiving and unable to discontinue medication which are strong inducers, strong inhibitors or enzyme substrates of cytochrome P450 CYP2C9 and CYP2C19 from 14 days prior to treatment.
8. Grade 3 bleeding symptoms (NCI-CTCAE v5.0) within 4 weeks prior to starting study treatment.
9. Unable to swallow IP or has refractory nausea and vomiting, malabsorption, external biliary diversion, or any significant small bowel resection that may interfere with adequate absorption of IP.
10. ECG QTcB≥480msec in screening, or history of congenital long QT syndrome.
11. Left ventricular ejection fraction (LVEF) <50%.
12. History major cerebrovascular diseases within 6 months prior to enrollment.
13. Infectious diseases requiring systemic treatment.
14. History or current evidence of retinal diseases.
15. Have active/chronic infection with hepatitis C, or positive hepatitis B surface antigen (HBsAg), or active/chronic infection with human immunodeficiency virus (HIV).
16. Known active tuberculosis.
17. History of allogeneic bone marrow transplantation or organ transplantation.
18. Interstitial lung disease or interstitial pneumonitis, including clinically significant radiation pneumonitis.
19. Pregnant or breast-feeding females.
20. Previous or history of second malignancy within 5 years prior to study treatment
21. Other conditions which may increase the risk associated with study participation, or interfere with the evaluation of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2020-11-12 (Actual); Study Completion 2020-11-12 (Actual)

PRIMARY OUTCOMES:
Adverse events (AEs) | Duration of the study, estimated to be approximately 24 months.
  An AE is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Dose limitation toxicities (DLT) | During Cycle 1 (the first 28 days)
  A DLT is defined as the occurrence of any of the following AE considered possibly, probably, or definitely related to the IP, HL-085, by the Investigator and/or the Sponsor that occurs during Cycle 1 as described in below:
  * Any death not clearly due to the underlying disease or extraneous causes; or
  * Non-hematologic toxicities Grade 3 or higher.
  * Grade 3 thrombocytopenia with clinically significant bleeding, or other hematologic toxicity at Grade 4 or above.
  * Neutropenic fever
  * liver parameter abnormalities
  * Any toxicity requiring permanent discontinuation of the IP
Maximum tolerated dose (MTD) | MTD will be determined when DLT occurs in great or equal to 33.3% of the same cohort subjects during During Cycle 1 (the first 28 days)
  MTD is defined as the highest dose level at which DLT occurs in less than 33.3% of subjects.

SECONDARY OUTCOMES:
cMAX | Duration of the study, estimated to be approximately 24 months
  cMAX is the maximum plasma concentration of HL-085 or metabolite(s).
Overall response rate (ORR) | Duration of the study, estimated to be approximately 24 months
  ORR is the proportion of patients with a best overall response of complete response (CR) or partial response (PR), as assessed per response evaluation criteria in solid tumors (RECIST) v1.1.

OTHER OUTCOMES:
pERK expression | Duration of the study, estimated to be approximately 24 months
  Correlation between phosphorylated extracellular-signal-regulated kinase (pERK) expression and efficacy endpoints.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Liu, MD, PhD, Study Director — KeChow Pharma
Locations (2):
- United States (2):
  - Livestrong Cancer Institute, Dell Medical School, The University of Texas at Austin, Austin, Texas
  - Next Oncology, San Antonio, Texas